CLINICAL TRIAL: NCT02848950
Title: The Effect of Metformin on Fecundability in Obese Women Undergoing ART - the Correlation to Uterine Flow Parameters A Prospective Randomized Controlled Trial
Brief Title: The Effect of Metformin on Fecundability in an ART(Assisted Reproductive Technology) Setting - the Correlation to Uterine Flows
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, nora gorhad, DOCTOR, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M.UTERUS.CTIL
Record Dates: First submitted 2016-05-17; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Infertility Female
Keywords: Metformin; fecundability; uterine doppler
MeSH Terms: conditions — Infertility, Female | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Active Comparator): drug: metformin
  Interventions: Drug: Metformin
- control (No Intervention): without metformin

INTERVENTIONS:
Drug: Metformin — Supplementation of the study group with Metformin till the day of pregnancy confirmation
  Other Names: glucophage
  Arms: treatment

SUMMARY:
The basis for obesity's impact on reproduction is not well characterised and there is a controversy whether the key organ influenced by it are the ovaries or the uterus.

Insulin sensitizers ameliorate insulin resistance in obese patients. This study seeks to determine if Metformin helps to increase fecundability by affecting the uterus in women undergoing ART. As a surrogate marker- flows in the uterus will be tested during the treatment.

DETAILED DESCRIPTION:
Obesity has been long implicated in reduced reproductive potential and it has been shown to impair conception and implantation. However, the basis for this adverse effect is still obscure and there is a controversy whether the key organ influenced by it are the ovaries or the uterus.

It is well established that insulin resistance is one of the main mechanisms of obesity's negative influences on the reproductive organs in females. Insulin sensitizers ameliorate insulin resistance in obese patients.

This study seeks to determine if Metformin ,an oral antidiabetic and insulin sensitizer, helps to increase fecundability by affecting the uterus in women undergoing frozen-thawed embryo transfer compared to the control group. As a surrogate marker- flows in the uterus will be tested during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18-40 years old.
* BMI > 30
* Infertile women undergoing frozen-thawed embryo transfer in an ART setting
* Women with at least one Top graded embryo
* Normal uterine Doppler indices at time of recruitment.

Exclusion Criteria:

* Diabetes mellitus - uncontrolled.
* Hyperprolactinemia- uncontrolled.
* Hypothyroidism- uncontrolled.
* women who are already treated with Metformin
* women with endometrial factor as the cause for infertility

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | until the blood test for pregnancy, about 4-6 weeks

SECONDARY OUTCOMES:
The changes in Doppler blood flow indices in both uterine arteries | until the blood test for pregnancy, about 4-6 weeks
endometrial thickness change measured by millimeters | until the blood test for pregnancy, about 4-6 weeks
Endometrial Doppler flows measured by power doppler - percentage of endometrium with flows | until the blood test for pregnancy, about 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JOHNNY YOUNIS, PEOFESSOR, Principal Investigator — Head of Fertility unit, Poriya' Bar Ilan University

IPD SHARING:
Plan to Share IPD: No